CLINICAL TRIAL: NCT02711800
Title: Probiotic Treatment: The Role of the Gut Microbiome in Childhood Abdominal Pain and Anxiety
Brief Title: The Probiotic Study: Using Bacteria to Calm Your Mind
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nancy Zucker (Other)
Responsible Party: Sponsor-Investigator, Nancy Zucker, Director of the Duke Center for Eating Disorders, Associate Professor in the Department of Psychology & Neuroscience, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00063870
Record Dates: First submitted 2016-01-22; First posted 2016-03-17 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Anxiety; Abdominal Pain
MeSH Terms: conditions — Anxiety Disorders; Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lactobacillus rhamnosus (Experimental): The investigators will use Culturelle®, a probiotic composed of the micro-organisms Lactobacillus GG. This formulation has been used for the treatment of gastrointestinal inflammation in numerous clinical trials. Dosing will follow the manufacturer's recommendation for children (1 capsule/packet per day), and will be monitored by Dr. Patrick Seed from the department of pediatrics. Weekly side effects and clinical changes will be monitored by both study therapist and caregiver using the Children's Global Assessment Scale and the Clinical Global Impression Scale (Severity, Improvement, and Efficacy). The intervention duration is 30 days.
  Interventions: Drug: Lactobacillus rhamnosus

INTERVENTIONS:
Drug: Lactobacillus rhamnosus — The investigators will use Culturelle®, a probiotic composed of the micro-organisms Lactobacillus GG. This formulation has been used for the treatment of gastrointestinal inflammation in numerous clinical trials. Dosing will follow the manufacturer's recommendation for children (1 capsule/packet per day), and will be monitored by the study Co-PI, Dr. Seed. Weekly side effects and clinical changes will be monitored by both study therapist and caregiver using the Children's Global Assessment Scale and the Clinical Global Impression Scale (Severity, Improvement, and Efficacy). The treatment duration is 30 days.
  Other Names: Culturelle Kids

SUMMARY:
The investigators seek to conduct the first open-label trial of probiotics in young children to reduce their anxiety and abdominal pain. Likewise, the investigators aim to assess the feasibility and efficacy of this treatment and to elucidate the enteric microbiota in the middle-lower GI tract. Self-report measures and a laboratory task will be collected from children, ages 9-13 years of age, and self-report measures from their primary caregivers prior to and following a 30-day probiotic administration. Children who score above cutoff in anxiety and/or abdominal pain meet the inclusion criteria for this study. Because of limited sample size and the iterative nature of intervention development, criteria for success at the pilot phase are based primarily on clinical rather than statistical criteria. The study personnel will do their best to keep and ensure the privacy and confidentiality of our participants; however, some of the risks of this study may include psychological discomfort, legal risks, and loss of confidentially.

ELIGIBILITY:
Inclusion Criteria:

Participants need to meet the criteria for functional abdominal pain as specified by the Rome III:

Scenario #1 Criteria for inclusion

1. In the last 2 months, how often did the child have pain or an uncomfortable feeling in the upper abdomen above the belly button? If ≥ 8 (or if the combination of #1 and #2 is ≥8)
2. In the last 2 months, how often did the child have pain or an uncomfortable feeling in the upper abdomen below the belly button? If ≥ 8 (or if the combination of #1 and #2 is ≥8)

Scenario #2 Criteria for inclusion 3. In the last 2 months, when the child hurt or felt uncomfortable above (below) the belly button, how often did your child miss school or stop activities? If #1 and #2 is ≥ 2 (or if the combination of #1 and #2 is ≥2) and #3 is ≥ 25% of the time.

They also have to be at or above cutoff (i.e. TS>= 55) for Beck Youth Inventory (BYI) which can be determined by finding the corresponding raw score, gender, and age on Appendix A in the BYI manual.

Exclusion Criteria:

1. Participants with immune disorders will be automatically excluded from this study.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Zucker, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke Center for Developmental Epedimiology, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Given the pilot nature of the study, resulting data may not be appropriate for sharing within a larger data repository. We will change this policy if we learn otherwise.

REFERENCES:
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159

RESULTS

PARTICIPANT FLOW:
Groups:
- Lactobacillus Rhamnosus: The investigators will use Culturelle®, a probiotic composed of the micro-organisms Lactobacillus GG. Dosing will follow the manufacturer's recommendation for children (1 capsule/packet per day), and will be monitored by Dr. Patrick Seed from the department of pediatrics. The intervention duration is 30 days.
Period: Overall Study
Arm/Group | Lactobacillus Rhamnosus
Started | 9
Completed | 7
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lactobacillus Rhamnosus
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.746 (0.753)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Pain intensity [Mean (Standard Deviation); unit: units on a scale] — Child and parent report is used to obtain ratings of pain intensity on a 0-12 scale. A lower score equates to lower pain intensity. Population: Data was missing for 3 participants
  units on a scale
    number analyzed (Participants) | 6
    (all) | 1.11 (1.04)

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Abdominal Pain Rating
Description: Child and parent report is used to obtain ratings of pain intensity on a 0-12 scale. A lower score equates to lower pain intensity. Ratings are obtained for a one-week period pre and post intervention, and measured 3 times daily. Pre-treatment assessments took place days 1-7, participants were treated days 8-36, and post-intervention assessments were completed days 37-44. All time points will be averaged and combined across raters (child and parent) resulting in an average pain severity rating pre and post-treatment. The change in this average rating will be assessed as pain severity outcome. This measure was averaged with the pain frequency average score (see Primary Outcome 2) to result in one primary severity/frequency pain rating pre and post treatment. The change in this combined measure is our primary index of change.
Time Frame: One week pre-intervention (Study Day 1), One week post-intervention (Study Day 44)
Population: Data was missing for one participant
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lactobacillus Rhamnosus
Number analyzed (Participants) | 6
units on a scale | 0.36 (0.58)

2. Primary Outcome: Change in Child Abdominal Pain Frequency
Description: Child and parent report is used to obtain ratings of pain frequency, the number of distinct occasions that pain was reported. Frequency was obtained for a one-week period pre and post intervention, and measured 3 times daily during these intervals. During the 30-day intervention, end of day frequencies were made. Pre-treatment assessments took place days 1-7, participants were treated days 8-36, and post-intervention assessments were completed days 37-44. The average number of episodes across these time points will be calculated pre and post treatment. The change in this average frequency from pre to post treatment will be the measure of change.
Time Frame: One week pre-intervention (Study Day 1), One week post-intervention (Study Day 44)
Population: Data was missing for one participant
Measure: Mean (Standard Deviation); unit: pain episodes
Arm/Group | Lactobacillus Rhamnosus
Number analyzed (Participants) | 6
pain episodes | 0.40 (0.61)

3. Primary Outcome: Change in Child Anxiety Symptoms
Description: We report the change in magnitude of self-reported state anxiety derived from summed raw scores obtained through the six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory at baseline and 30 days from baseline. Scores in the scale range from 6-24, with greater scores indicating worse anxiety. We obtained the summed raw scores after reverse scoring items 1, 4 & 5.
Time Frame: Baseline and 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lactobacillus Rhamnosus
Number analyzed (Participants) | 7
units on a scale | 1.30 (3.91)

4. Secondary Outcome: Percentage of Adherence to Treatment
Description: Adherence was calculated as: ("the days probiotic was taken"/"total number of days of treatment") x 100, with results ranging from 0% (no probiotics taken at all) to 100% (probiotics taken 30 days out of the 30 day-treatment period). Researcher will subtract the number of pills/packets taken from the total amount.
Time Frame: 30 days
Measure: Mean (Full Range); unit: percentage of adherence
Arm/Group | Lactobacillus Rhamnosus
Number analyzed (Participants) | 7
percentage of adherence | 91 [77 to 100]

5. Secondary Outcome: Change in Relative Quantities of Taxa Among Groups Relative to Probiotic Administration
Time Frame: Baseline and 30 days
Reporting Status: Not Posted, anticipated posting 2019-04

6. Secondary Outcome: Change in Alpha Diversity
Time Frame: Baseline and 30 days
Reporting Status: Not Posted, anticipated posting 2019-04

7. Secondary Outcome: Change in Beta Diversity (PCoA)
Time Frame: Baseline and 30 days
Reporting Status: Not Posted, anticipated posting 2019-04

8. Secondary Outcome: Change in Trait-associated Co-functional Modules of Organisms
Time Frame: Baseline and 30 days
Reporting Status: Not Posted, anticipated posting 2019-04

9. Secondary Outcome: Change in Salivary Cortisol (ug/dL)
Time Frame: Baseline and 30 days
Population: Three participants excluded from analysis: 2 with no post-treatment data, 1 with neither pre- nor post-treatment data.
Measure: Mean (Standard Deviation); unit: ug/dl
Arm/Group | Lactobacillus Rhamnosus
Number analyzed (Participants) | 6
ug/dl | -0.02 (0.06)

10. Secondary Outcome: Change in Heart Rate
Description: Beats per minute (Bpm)
Time Frame: Baseline and 30 days
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Lactobacillus Rhamnosus
Number analyzed (Participants) | 7
Beats per minute | 0.825 (6.056)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Lactobacillus Rhamnosus
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-07-31): https://cdn.clinicaltrials.gov/large-docs/00/NCT02711800/Prot_SAP_000.pdf